CLINICAL TRIAL: NCT04989504
Title: Mepitel Film for the Reduction of Radiation Dermatitis in Breast Cancer Patients Undergoing Post-Mastectomy Radiation Therapy: A Randomized Phase III Clinical Trial
Brief Title: Testing the Application of Mepitel Film During Radiation Therapy to Reduce Radiation Related Redness and Peeling in Breast Cancer Patients Following Mastectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A221803; NCI-2019-04688 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Carcinoma; Mastectomy Patient
MeSH Terms: conditions — Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Bandages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients receive standard of care skin management during radiation therapy for up to 6 weeks.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Mepitel Film) (Experimental): Patients receive Mepitel Film applied to breast or chest wall every week before radiation therapy for up to 6 weeks.
  Interventions: Device: Wound Dressing Material; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: Standard of Care
  Arms: Arm I (standard of care)
Device: Wound Dressing Material — Apply Mepitel Film
  Arms: Arm II (Mepitel Film)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well Mepitel Film works in reducing radiation dermatitis (redness and peeling) in patients with breast cancer during radiation therapy after a mastectomy. Mepitel Film may reduce the severity of skin redness and peeling in the area of radiation.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To determine the ability of Mepitel Film to reduce the severity of radiation dermatitis in patients undergoing post-mastectomy radiotherapy for breast cancer when compared to the institutional standard of care.

KEY SECONDARY OBJECTIVES:

I. To determine the ability of Mepitel Film to prevent radiation-induced dermatitis based on a centralized, blinded provider assessment review of photographs.

II. To determine the ability of Mepitel Film to prevent radiation-induced dermatitis based on a non-blinded institutional provider assessment.

III. To determine the ability of Mepitel Film to prevent radiation-induced dermatitis based on a combined patient and non-blinded institutional provider assessment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care skin management during radiation therapy for up to 6 weeks.

ARM II: Patients receive Mepitel Film applied to breast or chest wall every week before radiation therapy for up to 6 weeks.

After completion of study, patients are followed up at 7-14 days, 3 months, 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of breast malignancy with TNM staging.
* Patients must have undergone a mastectomy with or without reconstruction within the past 120 days if not receiving adjuvant therapy, or within 60 days after completion of the last dose of chemotherapy.
* No prior radiotherapy to any portion of the planned treatment site.
* No documented history of adhesive or tape allergy.
* Patients must be scheduled to receive conventionally fractionated photon-based radiation. Patients planning brachytherapy within the treatment field, and patients scheduled to receive bilateral radiation or hypofractionated radiation are not eligible.
* No active rash or pre-existing dermatitis within the treatment field.
* No co-existing medical conditions resulting in life expectancy < 2 years.
* No active collagen vascular diseases (i.e. lupus erythematosus, scleroderma, dermatomyositis).
* No concomitant cytotoxic chemotherapy. Endocrine therapy and HER2 directed therapies are allowed.
* No current inflammatory breast cancer, or gross dermal involvement at initiation of radiotherapy.
* No previous history of organ or bone marrow transplant.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* In order to complete the mandatory patient-completed measures, participants must be able to speak and read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2029-02-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Corbin, MD, Study Chair — Mayo Clinic
Locations (49):
- United States (49):
  - Fremont - Rideout Cancer Center, Marysville, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Glens Falls Hospital, Glens Falls, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Altru Cancer Center, Grand Forks, North Dakota
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - MUSC Health Tidelands Health Radiation Therapy Center, Murrells Inlet, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Doctor's Hospital of Laredo, Laredo, Texas
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Standard of Care): Patients receive standard of care skin management during radiation therapy for up to 6 weeks.>
  > Best Practice: Receive standard of care>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Arm II (Mepitel Film): Patients receive Mepitel Film applied to breast or chest wall every week before radiation therapy for up to 6 weeks.>
  > Wound Dressing Material: Apply Mepitel Film>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Standard of Care) | Arm II (Mepitel Film)
Started | 73 | 143
Completed | 65 | 143
Not Completed | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard of Care) | Arm II (Mepitel Film) | Total
Number analyzed (Participants) | 73 | 143 | 216
Age, Continuous [Median (Full Range); unit: years] | 53 [26 to 91] | 53 [25 to 87] | 53 [25 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 142 | 213
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 66 | 129 | 195
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 14 | 25
  White | 58 | 123 | 181
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 4 | 5
Ever Received Boost [Count of Participants; unit: Participants]
  Yes | 20 | 27 | 47
  No | 53 | 116 | 169

OUTCOME MEASURES:

1. Primary Outcome: Serially Measured Patient-completed Modified Radiation Induced Skin Reaction Assessment Scale (mRISRAS) Scores
Description: Scores obtained at baseline (i.e. prior to the start of radiation), during weekly radiation therapy, at 10 (±4) days post-radiation therapy, and at 3-months post radiation therapy. At a given measurement time point, a patient-completed mRISRAS score ranges from 0 to 12, where higher scores correspond to increased radiation-induced skin reactions. The effect of the Mepitel Film in reducing the severity of radiation dermatitis will be defined as the between-arm difference in the summary statistic area under the curve obtained from a repeated-measures (means) mixed model.
Time Frame: Up to 5 months
Measure: Median (95% Confidence Interval); unit: score on a scale*month
Groups:
- Arm I (Standard of Care): Patients receive standard of care skin management during radiation therapy for up to 6 weeks.
  >
  > Best Practice: Receive standard of care
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- Arm II (Mepitel Film): Patients receive Mepitel Film applied to breast or chest wall every week before radiation therapy for up to 6 weeks.
  >
  > Wound Dressing Material: Apply Mepitel Film
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
Arm/Group | Arm I (Standard of Care) | Arm II (Mepitel Film)
Number analyzed (Participants) | 60 | 132
score on a scale*month | 46.24 [38.42 to 54.06] | 35.32 [29.40 to 41.23]

2. Secondary Outcome: Centralized, Blinded Provider-completed Modified Radiation Induced Skin Reaction Assessment Scale (mRISRAS) Scores Obtained From a Blinded Grading of the Photographs Taken at the End of Radiation Therapy
Description: At the completion of radiation therapy, photographs will be obtained one hour after the removal of the Mepitel Film or immediately following completion of radiation therapy for patients on the standard of care arm. A panel of radiation oncology providers will perform the blinded, central review to score the photographs. Each provider will independently assign a provider-completed mRISRAS score to each photograph, and the average score will be calculated for each patient. The provider-completed mRISRAS score ranges from 0 to 24, where higher scores correspond to increased radiation-induced skin reactions. The Wilcoxon rank-sum test will be used to test for an effect of the Mepitel Film.
Time Frame: Up to 2 months
Reporting Status: Not Posted

3. Secondary Outcome: Serially Measured Non-blinded Institutional Provider-completed Modified Radiation Induced Skin Reaction Assessment Scale (mRISRAS) Scores
Description: Scores obtained at baseline (i.e. prior to the start of radiation), during weekly radiation therapy, at 10 (±4) days post-radiation therapy, and at 3-months post radiation therapy. At a given measurement time point, a provider-completed mRISRAS score ranges from 0 to 24, where higher scores correspond to increased radiation-induced skin reactions. The effect of the Mepitel Film in reducing the severity of radiation dermatitis will be defined as the between-arm difference in the summary statistic area under the curve obtained from a repeated-measures (means) mixed model.
Time Frame: Up to 5 months
Measure: Median (Full Range); unit: score on a scale*month
Arm/Group | Arm I (Standard of Care) | Arm II (Mepitel Film)
Number analyzed (Participants) | 60 | 132
score on a scale*month | 8.0 [7.0 to 9.0] | 8.0 [3.0 to 9.0]

4. Secondary Outcome: Serially Measured Combined Patient- and Provider-completed Modified Radiation Induced Skin Reaction Assessment Scale (mRISRAS) Scores
Description: Scores obtained at baseline (i.e. prior to the start of radiation), during weekly radiation therapy, at 10 (±4) days post-radiation therapy, and at 3-months post radiation therapy. At a given measurement time point, a provider-completed mRISRAS score ranges from 0 to 36, where higher scores correspond to increased radiation-induced skin reactions. The effect of the Mepitel Film in reducing the severity of radiation dermatitis will be defined as the between-arm difference in the summary statistic area under the curve obtained from a repeated-measures (means) mixed model.
Time Frame: Up to 5 months
Measure: Median (Full Range); unit: score on a scale*month
Arm/Group | Arm I (Standard of Care) | Arm II (Mepitel Film)
Number analyzed (Participants) | 60 | 132
score on a scale*month | 16.0 [14.0 to 18.0] | 16.0 [6.0 to 18.0]

ADVERSE EVENTS:
Time Frame: Up to 5 months
Arm/Group | Arm I (Standard of Care) | Arm II (Mepitel Film)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/143
Serious Adverse Events (participants affected / at risk) | 2/65 | 7/143
Other Adverse Events (participants affected / at risk) | 59/65 | 133/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Standard of Care) (N=65) | Arm II (Mepitel Film) (N=143)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Standard of Care) (N=65) | Arm II (Mepitel Film) (N=143)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (6)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 8 (20)
Nausea (Gastrointestinal disorders) | 8 (18) | 8 (18)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 18 (58) | 33 (80)
Fever (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 3 (10) | 9 (22)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 5 (10)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 2 (3)
Shingles (Infections and infestations) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 8 (14)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 56 (211) | 115 (351)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (10)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (5)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 1 (4) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 4 (5)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 4 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (8) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (8) | 0 (0)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 3 (7) | 3 (3)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5) | 3 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (6)
Chronic kidney disease (Renal and urinary disorders) | 1 (6) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 9 (26) | 8 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (12) | 3 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (24)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 4 (9) | 3 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 44 (128) | 99 (306)
Rash acneiform (Skin and subcutaneous tissue disorders) | 15 (30) | 30 (64)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (18) | 21 (43)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (23)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 4 (15) | 2 (4)
Hypertension (Vascular disorders) | 5 (20) | 5 (11)
Lymphedema (Vascular disorders) | 1 (5) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 1 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT04989504/Prot_SAP_000.pdf